CLINICAL TRIAL: NCT04571450
Title: Effects On Blood Pressure And Body Composition Of A Self-Applied Online Re-Intervention Focused On Healthy Eating And Increased Physical Activity On Hypertensive Adults With Overweight Or Obesity.
Brief Title: Lifestyle Online Re-Intervention On Blood Pressure, BMI, And Physical Activity On Obese Hypertensive Patients
Acronym: IBI-HTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Professor of the Deparment of Biomedical Sciences, Cardenal Herrera University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-26
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Hypertension; Overweight and Obesity
Keywords: Hypertension; Obesity; Internet; Exercise; Nutrition; Reintervention
MeSH Terms: conditions — Hypertension; Overweight; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): All participants will receive access to the same web-based lifestyle intervention (exercise and nutritional education)
  Interventions: Behavioral: Reintervention

INTERVENTIONS:
Behavioral: Reintervention — This self-applied online program will take three months and comprise 9 behavioural modules developed gradually, achieving the changes needed on eating and physical activity habits, supported by audiovisual instructions given by an hypertension specialist doctor.

SUMMARY:
This research will constitute a 3 years follow-up which includes a re-assessment and re-intervention of obese or overweight adults with hypertension, recruited from a hypertension unit of a public hospital, that already participated in a similar program 3 years ago. At the same time, the aim of the study is to analyze the effects of the current program, which will take 3 months and promotes lifestyle changes focusing on healthy eating and increased physical activity in their 9 modules, comparing the results obtained in 2018. These patients will be allocated into one experimental group. Assessment will include: Blood Pressure, Body Mass Index, Physical Activity levels, and adherence to the Mediterranean diet.

DETAILED DESCRIPTION:
Hypertension incidence and overweight or obesity related, constitute a worrying public health problem nowadays. In this sense, healthy eating and regular physical activity have demonstrated a relevant role maintaining health while ageing. Information and Communication Technologies (ICTs) have been shown as a useful way to promote health, improving motivation and overcoming difficulties to maintain a healthy lifestyle. ICTs also reach a wider audience at a lower cost, due to their good cost-benefit relationship and the possibility of increasing the efficiency of interventions.

This research will constitute a 3 years follow-up which includes a re-assessment and re-intervention of obese or overweight adults with hypertension, recruited from a hypertension unit of a public hospital, that already participated in a similar program 3 years ago. At the same time, the aim of the study is to analyze the effects of the current program, which will take 3 months and promotes lifestyle changes focusing on healthy eating and increased physical activity in their 9 modules, comparing the results obtained in 2018. These patients will be allocated into one experimental group. Assessment will include: Blood Pressure, Body Mass Index, Physical Activity levels, and adherence to the Mediterranean diet.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension
* Overweight or obesity (25 ≤ BMI ≤ 35 kg/m2)
* Aged between 18-65 years
* Have participated in the same program 3 years ago

Exclusion Criteria:

* Not having access to the Internet or lack of information about it.
* Treatment with more than 3 antihypertensive drugs.
* Meet the criteria of the DSM-IV-TR of a Food Disorder.
* Presenting some type of severe psychiatric disorder.
* Disability that prevents or hinders physical exercise.
* Receiving some treatment for weight loss.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Blood Pressure (BP) | 3 months
  Systolic and diastolic blood pressure

SECONDARY OUTCOMES:
BMI | 3 months
  Body Mass Index
Physical activity | 3 months
  Levels of physical activity (measured with SHORT-IPAQ Questionnaire). This Questionnaire assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.

CONTACTS AND LOCATIONS:
Overall Officials: JUAN FRANCISCO L Lisón Párraga, PhD, Principal Investigator — Cardenal Herrera University
Locations (1):
- Juan Francisco Lisón Párraga, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lison JF, Palomar G, Mensorio MS, Banos RM, Cebolla-Marti A, Botella C, Benavent-Caballer V, Rodilla E. Impact of a Web-Based Exercise and Nutritional Education Intervention in Patients Who Are Obese With Hypertension: Randomized Wait-List Controlled Trial. J Med Internet Res. 2020 Apr 14;22(4):e14196. doi: 10.2196/14196. PMID 32286232